CLINICAL TRIAL: NCT04096326
Title: A Phase 2b Double-Blind, Placebo-Controlled, Dose-Ranging Study to Evaluate the Safety and Efficacy of AGN-151586 in Participants With Moderate to Severe Glabellar Lines
Brief Title: AGN-151586 Dose-Ranging Study for Treatment of Glabellar Lines
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2034-201-008
Record Dates: First submitted 2019-09-04; First posted 2019-09-19 (Actual); Results first posted 2023-07-28 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Glabellar Lines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (10):
- Cohort 1: Placebo (Placebo Comparator): Participants received AGN-151586-matching placebo, intramuscular (IM) injections in the glabellar complex on Day 1 in Cohort 1.
  Interventions: Drug: Placebo
- Cohort 1: AGN-151586 (Experimental): Participants received AGN-151586 lowest dose, IM injections in the glabellar complex on Day 1.
  Interventions: Drug: AGN-151586
- Cohort 2: Placebo (Placebo Comparator): Participants received AGN-151586-matching placebo, IM injections in the glabellar complex on Day 1 in Cohort 2.
  Interventions: Drug: Placebo
- Cohort 2: AGN-151586 (Experimental): Participants received AGN-151586, IM injections in the glabellar complex on Day 1.
  Interventions: Drug: AGN-151586
- Cohort 3: Placebo (Placebo Comparator): Participants received AGN-151586-matching placebo, IM injections in the glabellar complex on Day 1 in Cohort 3.
  Interventions: Drug: Placebo
- Cohort 3: AGN-151586 (Experimental): Participants received AGN-151586, IM injections in the glabellar complex on Day 1.
  Interventions: Drug: AGN-151586
- Cohort 4: Placebo (Placebo Comparator): Participants received AGN-151586-matching placebo, IM injections in the glabellar complex on Day 1 in Cohort 4.
  Interventions: Drug: Placebo
- Cohort 4: AGN-151586 (Experimental): Participants received AGN-151586, IM injections in the glabellar complex on Day 1.
  Interventions: Drug: AGN-151586
- Cohort 5: Placebo (Placebo Comparator): Participants received AGN-151586-matching placebo, IM injections in the glabellar complex on Day 1 in Cohort 5.
  Interventions: Drug: Placebo
- Cohort 5: AGN-151586 (Experimental): Participants received AGN-151586 highest dose, IM injections in the glabellar complex on Day 1.
  Interventions: Drug: AGN-151586

INTERVENTIONS:
Drug: AGN-151586 — AGN-151586 solution for injection.
  Arms: Cohort 1: AGN-151586; Cohort 2: AGN-151586; Cohort 3: AGN-151586; Cohort 4: AGN-151586; Cohort 5: AGN-151586
Drug: Placebo — Placebo solution for injection.
  Arms: Cohort 1: Placebo; Cohort 2: Placebo; Cohort 3: Placebo; Cohort 4: Placebo; Cohort 5: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of AGN-151586 over a range of doses for the treatment of moderate to severe glabellar lines (GL).

ELIGIBILITY:
Inclusion Criteria:

-Female participants willing to minimize the risk of inducing pregnancy for the duration of the clinical study and follow-up period (at least 10 weeks after study intervention).

Exclusion Criteria:

* Known immunization or hypersensitivity to any botulinum neurotoxin serotype
* Any medical condition that may put the participant at increased risk with exposure to AGN-151586, including diagnosed myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis, or any other condition that might interfere with neuromuscular function
* Marked facial asymmetry, dermatochalasis, deep dermal scarring, excessively thick sebaceous skin, or the inability to substantially lessen facial lines even by physically spreading them apart, as determined by the investigator
* Any brow or eyelid ptosis, as determined by the investigator
* Infection or skin disorder at the injection sites
* History of facial nerve palsy
* Any uncontrolled systemic disease
* Anticipated need for treatment with botulinum neurotoxin of any serotype for any reason during the study (other than study intervention)
* Anticipated need for surgery or overnight hospitalization during the study
* Prior periorbital surgery, facial lift (full face or mid-face), thread lift, brow lift, or related procedures (eg, eyelid [blepharoplasty] and/or eyebrow surgery)
* Prior facial treatment with permanent soft tissue fillers, synthetic implantation (eg, Gore-Tex®), and/or autologous fat transplantation
* Current enrollment in an investigational drug or device study or participation in such a study within 30 days of Screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2019-09-26 (Actual); Primary Completion 2020-09-09 (Actual); Study Completion 2020-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ALLERGAN INC., Study Director — Allergan
Locations (9):
- United States (9):
  - Center for Dermatology Clinical Research /ID# 237798, Fremont, California
  - Ava T. Shamban MD - Santa Monica. /ID# 235353, Santa Monica, California
  - Skin and Cancer Associates, LLP /ID# 236231, Miami, Florida
  - Laser and Skin Surgery Center of Indiana /ID# 236588, Indianapolis, Indiana
  - Wilmington Dermatology Center /ID# 237055, Wilmington, North Carolina
  - Kgl, Llc /Id# 234798, Newtown Square, Pennsylvania
  - DermResearch Inc. /ID# 234483, Austin, Texas
  - Austin Institute for Clinical Research at SBA Dermatology /ID# 236646, Houston, Texas
  - Austin Institute for Clinical Research /ID# 237135, Pflugerville, Texas

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Additional information on study locations near you may be found at AllerganClinicalTrials.com. For any study not on AllerganClinicalTrials.com, please contact IR-CTRegistration@Allergan.com for assistance — http://www.AllerganClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 198 participants with moderate to severe glabellar lines (GL) were enrolled and randomized in a 3:1 ratio to receive AGN-151586 in 5 sequential AGN-151586 dose rising cohorts or Placebo in each of the 5 cohorts.
Period: Overall Study
Arm/Group | Cohort 1: Placebo | Cohort 1: AGN-151586 | Cohort 2: Placebo | Cohort 2: AGN-151586 | Cohort 3: Placebo | Cohort 3: AGN-151586 | Cohort 4: Placebo | Cohort 4: AGN-151586 | Cohort 5: Placebo | Cohort 5: AGN-151586
Started | 8 | 32 | 12 | 28 | 11 | 27 | 10 | 30 | 9 | 31
Completed | 8 | 31 | 12 | 28 | 10 | 22 | 9 | 30 | 9 | 31
Not Completed | 0 | 1 | 0 | 0 | 1 | 5 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — COVID-19-related reasons | 0 | 0 | 0 | 0 | 1 | 5 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Modified intent-to-treat (mITT) population included all randomized participants who received the study intervention and who had at least one postintervention investigator-rated facial wrinkle scale with photonumeric guide (FWS) measurement at maximum frown.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Placebo | Cohort 1: AGN-151586 | Cohort 2: Placebo | Cohort 2: AGN-151586 | Cohort 3: Placebo | Cohort 3: AGN-151586 | Cohort 4: Placebo | Cohort 4: AGN-151586 | Cohort 5: Placebo | Cohort 5: AGN-151586 | Total
Number analyzed (Participants) | 8 | 32 | 12 | 28 | 11 | 27 | 10 | 30 | 9 | 31 | 198
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.9 (6.24) | 52.8 (8.85) | 47.0 (9.39) | 50.9 (10.10) | 50.1 (10.63) | 47.5 (10.53) | 39.0 (7.94) | 45.3 (8.06) | 51.1 (11.37) | 46.4 (10.30) | 48.3 (9.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 29 | 12 | 25 | 11 | 24 | 9 | 26 | 9 | 30 | 182
  Male | 1 | 3 | 0 | 3 | 0 | 3 | 1 | 4 | 0 | 1 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 9 | 3 | 4 | 4 | 8 | 3 | 12 | 0 | 7 | 52
  Not Hispanic or Latino | 6 | 23 | 9 | 24 | 7 | 19 | 7 | 18 | 9 | 24 | 146
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 3 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 4
  Black or African American | 1 | 2 | 0 | 2 | 0 | 0 | 0 | 2 | 1 | 2 | 10
  White | 7 | 27 | 10 | 24 | 10 | 26 | 10 | 28 | 7 | 26 | 175
  More than one race | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With ≥ 2-grade Improvement From Baseline on the FWS According to Investigator's Assessment at Any Postintervention Timepoint Through Day 7
Description: Percentage of participants achieving a ≥ 2-grade improvement from baseline on the FWS according to investigator assessments of GL severity at maximum frown at any postintervention timepoint through Day 7 were reported. Investigators' assessments of the severity of GL at rest and maximum frown using the validated FWS was assessed using the 4-grade FWS, where 0=none, 1=mild, 2=moderate, and 3=severe. Higher scores indicate more severity. Percentages are rounded off to nearest single decimal.
Time Frame: Baseline (Day 1) through Day 7
Population: mITT population included all randomized participants who received the study intervention and who had at least one postintervention investigator-rated FWS measurement at maximum frown.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: Placebo | Cohort 1: AGN-151586 | Cohort 2: Placebo | Cohort 2: AGN-151586 | Cohort 3: Placebo | Cohort 3: AGN-151586 | Cohort 4: Placebo | Cohort 4: AGN-151586 | Cohort 5: Placebo | Cohort 5: AGN-151586
Number analyzed (Participants) | 8 | 32 | 12 | 28 | 11 | 27 | 10 | 30 | 9 | 31
percentage of participants | 0.0 [NA to NA] — Upper and lower limit of 95% CI was not estimable as there was no participant with response having at least ≥ 2-grade improvement from baseline at any postintervention timepoint through Day 7. | 40.6 [23.7 to 59.4] | 0.0 [NA to NA] — Upper and lower limit of 95% CI was not estimable as there was no participant with response having at least ≥ 2-grade improvement from baseline at any postintervention timepoint through Day 7. | 46.4 [27.5 to 66.1] | 18.2 [2.3 to 51.8] | 70.4 [49.8 to 86.2] | 20.0 [2.5 to 55.6] | 83.3 [65.3 to 94.4] | 11.1 [0.3 to 48.2] | 96.8 [83.3 to 99.9]
Statistical Analysis 1: Comparison: Cohort 1: Placebo vs Cohort 1: AGN-151586; Test type: Superiority; p = 0.0096, Cochran-Mantel-Haenszel — P-value was based on Cochran-Mantel-Haenszel (CMH) tests stratified by baseline GL severity at maximum frown to compare each AGN-151586 study intervention group versus placebo for each cohort; Rate difference = 40.6, 95% CI 2-sided [23.6 to 57.6]
Statistical Analysis 2: Comparison: Cohort 2: Placebo vs Cohort 2: AGN-151586; Test type: Superiority; p = 0.0094, Cochran-Mantel-Haenszel — P-value was based on CMH tests stratified by baseline GL severity at maximum frown to compare each AGN-151586 study intervention group versus placebo for each cohort; Rate difference = 46.4, 95% CI 2-sided [28.0 to 64.9]
Statistical Analysis 3: Comparison: Cohort 3: Placebo vs Cohort 3: AGN-151586; Test type: Superiority; p = 0.0044, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Rate difference = 52.2, 95% CI 2-sided [23.6 to 80.8]
Statistical Analysis 4: Comparison: Cohort 4: Placebo vs Cohort 4: AGN-151586; Test type: Superiority; p = 0.0026, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Rate difference = 63.3, 95% CI 2-sided [35.2 to 91.5]
Statistical Analysis 5: Comparison: Cohort 5: Placebo vs Cohort 5: AGN-151586; Test type: Superiority; p = 0.0000, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Rate difference = 85.7, 95% CI 2-sided [64.2 to 100.0]

2. Primary Outcome: Number of Participants Who Experience One or More Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study intervention, whether considered related to the study intervention or not. TEAEs were defined as events event began on or after the date and time of the study intervention; or the adverse event was present before the date and time of the study intervention, but increased in severity or became serious on or after the date and time of the study intervention.
Time Frame: From first dose of study drug until the end of study (up to 42 days)
Population: Safety population included all participants who received study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Placebo | Cohort 1: AGN-151586 | Cohort 2: Placebo | Cohort 2: AGN-151586 | Cohort 3: Placebo | Cohort 3: AGN-151586 | Cohort 4: Placebo | Cohort 4: AGN-151586 | Cohort 5: Placebo | Cohort 5: AGN-151586
Number analyzed (Participants) | 8 | 32 | 12 | 28 | 11 | 27 | 10 | 30 | 9 | 31
Participants | 3 | 15 | 7 | 10 | 7 | 9 | 3 | 9 | 1 | 12

3. Primary Outcome: Number of Participants With Potentially Clinically Significant Laboratory Parameters Post Intervention
Description: Potentially clinically significant post intervention laboratory values included hematology, chemistry, and urinalysis as defined in the SAP.
Time Frame: From first dose of study drug until the end of study (up to 42 days)
Population: Safety population included all participants who received study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Placebo | Cohort 1: AGN-151586 | Cohort 2: Placebo | Cohort 2: AGN-151586 | Cohort 3: Placebo | Cohort 3: AGN-151586 | Cohort 4: Placebo | Cohort 4: AGN-151586 | Cohort 5: Placebo | Cohort 5: AGN-151586
Number analyzed (Participants) | 8 | 32 | 12 | 28 | 11 | 27 | 10 | 30 | 9 | 31
Participants | 0 | 7 | 1 | 5 | 3 | 4 | 0 | 4 | 5 | 8

4. Primary Outcome: Number of Participants With Potentially Clinically Significant Vital Signs Post Intervention
Description: Potentially clinically significant post intervention vital sign measurements included systolic and diastolic blood pressure, pulse rate, respiration rate, body temperature as defined in the SAP.
Time Frame: From first dose of study drug until the end of study (up to 42 days)
Population: Safety population included all participants who received study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Placebo | Cohort 1: AGN-151586 | Cohort 2: Placebo | Cohort 2: AGN-151586 | Cohort 3: Placebo | Cohort 3: AGN-151586 | Cohort 4: Placebo | Cohort 4: AGN-151586 | Cohort 5: Placebo | Cohort 5: AGN-151586
Number analyzed (Participants) | 8 | 32 | 12 | 28 | 11 | 27 | 10 | 30 | 9 | 31
Participants | 2 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 1

5. Primary Outcome: Number of Participants With Potentially Clinically Significant Electrocardiogram Findings Post Intervention
Description: Potentially clinically significant post intervention values in 12-lead ECG recordings included heart rate and measures PR, QRS, QT and QTcF intervals. 12-lead ECG recordings were obtained after the participants have rested for at least 10 minutes in semi-supine or supine position as defined in the SAP. A post-baseline value is considered potentially clinically significant if it meets either the observed-value or the change-from-baseline criteria such as QRS interval observed value: ≥ 150 msec; PR interval observed value: ≥ 250 msec; QTcB observed value: > 500 msec or change from baseline value: increase of > 60 msec; QTcF observed value: > 500 msec or change from baseline value: increase of > 60 msec.
Time Frame: From first dose of study drug until the end of study (up to 42 days)
Population: Safety population included all participants who received study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Placebo | Cohort 1: AGN-151586 | Cohort 2: Placebo | Cohort 2: AGN-151586 | Cohort 3: Placebo | Cohort 3: AGN-151586 | Cohort 4: Placebo | Cohort 4: AGN-151586 | Cohort 5: Placebo | Cohort 5: AGN-151586
Number analyzed (Participants) | 8 | 32 | 12 | 28 | 11 | 27 | 10 | 30 | 9 | 31
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Number of Participants With Anti-drug Antibodies (ADAs)
Description: Number of participants with positive anti-drug antibodies are reported. Binding and neutralizing anti-bodies are evaluated as anti-drug antibodies. Only participants with positive samples for binding antibodies have been analyzed for presence of neutralizing antibodies.
Time Frame: Up to Day 42
Population: Safety population included all participants who received study intervention. Overall number of participants analyzed are the number of participants available for analyses. Number analyzed indicates the number of participants with data available for analysis for the below categories.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Placebo | Cohort 1: AGN-151586 | Cohort 2: Placebo | Cohort 2: AGN-151586 | Cohort 3: Placebo | Cohort 3: AGN-151586 | Cohort 4: Placebo | Cohort 4: AGN-151586 | Cohort 5: Placebo | Cohort 5: AGN-151586
Number analyzed (Participants) | 0 | 32 | 0 | 28 | 0 | 26 | 1 | 30 | 0 | 31
Participants
  Binding Antibodies | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Neutralizing Antibodies: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Neutralizing Antibodies | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality was reported from enrollment to the end of study; median time on follow-up was 42 days for the placebo and AGN-151586 arms, respectively. Treatment-emergent adverse events and serious adverse events were collected from first dose of study drug until 42 days after the last dose of study drug.
Description: Safety population included all participants who received study intervention.
Arm/Group | Cohort 1: Placebo | Cohort 1: AGN-151586 | Cohort 2: Placebo | Cohort 2: AGN-151586 | Cohort 3: Placebo | Cohort 3: AGN-151586 | Cohort 4: Placebo | Cohort 4: AGN-151586 | Cohort 5: Placebo | Cohort 5: AGN-151586
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/32 | 0/12 | 0/28 | 0/11 | 0/27 | 0/10 | 0/30 | 0/9 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/32 | 0/12 | 0/28 | 0/11 | 0/27 | 0/10 | 0/30 | 0/9 | 0/31
Other Adverse Events (participants affected / at risk) | 3/8 | 15/32 | 7/12 | 10/28 | 7/11 | 9/27 | 3/10 | 9/30 | 1/9 | 12/31
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Placebo (N=8) | Cohort 1: AGN-151586 (N=32) | Cohort 2: Placebo (N=12) | Cohort 2: AGN-151586 (N=28) | Cohort 3: Placebo (N=11) | Cohort 3: AGN-151586 (N=27) | Cohort 4: Placebo (N=10) | Cohort 4: AGN-151586 (N=30) | Cohort 5: Placebo (N=9) | Cohort 5: AGN-151586 (N=31)
Injection site pain (General disorders) | 0 | 6 | 3 | 1 | 1 | 7 | 2 | 4 | 0 | 6
Facial pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Chills (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site discomfort (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site haemorrhage (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site pruritus (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 2 | 2 | 4 | 2 | 1 | 3 | 2 | 0 | 2
Presyncope (Nervous system disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asymptomatic COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pharyngeal hypoaesthesia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Photophobia (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Stress (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Allergy to arthropod bite (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Breast induration (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-05-20): https://cdn.clinicaltrials.gov/large-docs/26/NCT04096326/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-13): https://cdn.clinicaltrials.gov/large-docs/26/NCT04096326/SAP_001.pdf